CLINICAL TRIAL: NCT06636032
Title: Dose Escalation of Allogeneic Adipose Derived Stroma/Stem Cells for the Treatment of Crohn's Fistula:a Phase I/II Clinical Study
Brief Title: Dose Escalation of Allogeneic Adipose Derived Stroma/Stem Cells for the Treatment of Crohn's Fistula
Acronym: ALLOFIST
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/13/7030
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease
Keywords: Crohn's disease; perianal fistula; regenerative medicine; immunomodulation; allogeneic adipose-derived stem cell
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AdMSC (CellReady®) (Experimental): Different doses of AdMSC will be tested for a dose escalation (5.10*7 and 10.10*7 cells) and injected in the in the wall of the fistula
  Interventions: Drug: AdMSC (CellReady®)

INTERVENTIONS:
Drug: AdMSC (CellReady®) — At day 0, patients will have AdMSC injections. Patients will be followed-up for 6 months
  Other Names: AdMSC

SUMMARY:
Perianal fistulas are in the forefront (42 to 72, 4%) of morbid complication of Crohn's disease, affecting nearly one- third of patients and complicating abscesses in 35-48% of cases. The current treatment is based on the combination of drainage (proctologic and surgical), and biologics techniques, but the failure rate varies from 30 to 80%. Actually, innovative cell therapy procedures are validated by Cell-Easy with the use of allogenic mesenchymal stem cells for the immunomodulatory, anti-inflammatory, angiogenic and trophic properties (CellReady®) and represent a promising option in the treatment of perianal fistulas associated with Crohn's disease. This phase I/II study is designed to evaluate the treatment of complex perianal fistulas associated with Crohn's disease, after failure of conventional treatment by injection of allogeneic cultured adipose-derived stromal cell (AdMSC) into the fistula.

DETAILED DESCRIPTION:
The injection of adipose stromal cells is currently evaluated in clinical studies for repair-damaged tissues in various diseases (limb ischemia, osteoarthritis, systemic slerosis...). Immunoregulatory and anti-inflammatory properties of AdMSC's are responsible for accelerating healing and represents an innovative approach to treat perianal fistulas associated with Crohn's disease.

This phase I/II study is designed to evaluate the treatment of complex perianal fistulas associated with Crohn's disease, after failure of conventional treatment by injection of AdMSC (CellReady®) into the fistula.

Different doses of AdMSC will be tested for a dose escalation (5.10*7 and 10.10*7 cells) and injected in the in the wall of the fistula.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old,
* Patients who signed the informed consent,
* Patient affiliated to a social security system,
* Controlled luminal Crohn's disease characterized by an Harvey-Bradshaw score less or equal than 8 and diagnosed on clinical, endoscopic, histological and/or radiological criteria for more than 3 months,
* Colonoscopy less than a year old without ulcer in the rectum,
* Presence of complex chronic perianal fistula with a maximum of two internal ports and three external ports,
* Patient treated with a combined treatment (drainage on setons + anti-TNFα) and who failed conventional treatment after 6 months and whose intraluminal disease (intestinal damage) is controlled

Exclusion Criteria:

* Refusal of the patient to participate in the study,
* Positive QuantiFERON test,
* Patient with transplanted organ,
* History of cancer in the last five years or lympho-proliferative disease,
* Persistent bacterial or viral infection,
* Patient with a contraindication to MRI,
* Known allergy to Gadolinium,
* Known allergy to Albumine,
* End-stage organ failure,
* Pregnant or breastfeeding women,
* Women of childbearing age without effective contraception throughout the duration of the study,
* Patient under judicial protection, under guardianship or curatorship.
* Patient previously treated with ALOFISEL®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
adverse events of grade ≥ 2 at 6 months | 6 months after injection
  Number of adverse events of grade ≥ 2 related to the experimental treatment (CellReady®) or related to surgical/medical procedures,
Efficacy of AdMSC by clinical evaluation at 6 months | 6 months after injection
  This evaluation will be measured by the presence or absence of flow through the internal or external orifice see in anoscopy and through the external orifice
Efficacy of AdMSC by radiological evaluation at 6 months | 6 months after injection
  This evaluation will be measured by disappearance of fistula tract or fistula tract present but inactive.

SECONDARY OUTCOMES:
Safety at 1 and 3 and 6 months | 1, 3 and 6 months after injection
  adverse effects will be assessed
Efficacy of AdMSC by clinical evaluation 1 and 3 months | 1 and 3 months after injection
  This evaluation will be measured by the presence or absence of flow through the internal or external orifice see in anoscopy and through the external orifice
Efficacy of AdMSC by biological evaluation | 1, 3 and 6 months after injection
  complete blood count , platelets, C-reactive protein (CRP) , liver enzyme profile, Prothrombin level (TP), activated clotting time (ACT), albumin, ferritinemia will be measured in blood samples
Change from Baseline in quality of life | 1, 3 and 6 months after injection
  Evaluation of quality of life by CAF QoL
Change from Baseline in disease activity | 1, 3 and 6 months after injection
  Evaluation of quality of life by Harvey-Bradshaw Index
Change from Baseline in perianal disease activity | 1, 3 and 6 months after injection
  Evaluation by perianal disease activity index (PDAI) . This index evaluate the presence of a fistula, the presence of pain and its impact on activity, the characteristics of the APL, the impact on the sexual activity
Change from Baseline in lesions | 1, 3 and 6 months after injection
  Evaluation by Cardiff classifcation . The creation of subclasses of anoperineal lesions allowing the comparison of superimposable groups in therapeutic trials. This classification allows a standardized and precise description of lesions.
Change from Baseline in anal incontinence | 1, 3 and 6 months after injection
  Evaluation by Wexner anal incontinence score: score to quickly and simply assess the severity of anal incontinence.
Change from Baseline in patient symptoms | 1, 3 and 6 months after injection
  Evaluation by Allan score: score used to assess patient symptoms and assess the impact of treatment on perineal lesions.
tryptophan metabolists | 3 and 6 months after injection
  tryptophan metabolists are measured by high pressure liquid chromatography coupled with tandem mass spectrometry
faecal microbiota | 3 and 6 months after injection
  faecal microbiota is analysed by Illumina Mi-Seq

CONTACTS AND LOCATIONS:
Overall Officials: Etienne BUSCAIL, MD, Principal Investigator — Toulouse Hospital
Locations (1):
- Toulouse Hospital, Toulouse, France

REFERENCES:
- [Derived] Buscail E, Gilletta de Saint Joseph C, Lebrin M, Frument I, Gross F, Bournet B, Buscail L, Culetto A, Mokrane F, Delchier MC, Quelven I, Daguzan C, Pugnet G, Duffas JP, Ghouti L, Philis A, Carrere N, Lepage B, Le Cosquer G. Rationale and design of the AlloFIST trial: a phase I/IIa study to evaluate dose escalation of allogeneic adipose-derived stroma/stem cells for the treatment of Crohn's fistula. BMJ Open. 2025 Dec 29;15(12):e104517. doi: 10.1136/bmjopen-2025-104517. PMID 41469061